CLINICAL TRIAL: NCT05443997
Title: To What Extent do Systems Strengthening Interventions and Engagement With Local Governance Improve the Quality and Co-coverage of Nutrition Services in Gujarat, India? A Cluster-randomized Evaluation
Brief Title: Systems Strengthening Interventions to Improve Quality and Co-coverage of Nutrition Services in Gujarat, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00007490
Record Dates: First submitted 2022-02-17; First posted 2022-07-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Maternal Nutrition
Keywords: Maternal Nutrition; Supportive supervision; MIYCN behaviors; System strengthening

STUDY DESIGN:
Intervention Model Description: The implementation research study uses a cluster-randomized design with cross-sectional baseline and endline surveys
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A&T- intensive (Experimental): 1. Capacity building will involve offsite training conducted by Vitamin Angels and short capsule trainings delivered by government staff
  2. Supportive supervision will involve training and handholding of supervisors on use of job aids and mobile application
  3. Strategic use of data will involve setting up processes to review key data, review meetings and short trainings on gap areas.
  4. Engagement of Panchayati Raj Institutions (PRI) around convergence where PRI members will be equipped with job aids, including an App
  5. Improved food supplements where THR offering for pregnant and lactating women and children 6 months and older will be revisited and improved solutions will be explored.
  Interventions: Behavioral: MIYCN capacity building
- A&T-non intensive (No Intervention): Only receives standard government services

INTERVENTIONS:
Behavioral: MIYCN capacity building — * MIYCN knowledge, skills, and motivation of FLWs
  * Supportive supervision
  * Decentralized programmatic decision-making using data
  * PRI member involvement
  * Availability of THR
  * IYCF knowledge and practices
  Other Names: Strengthening Supportive Supervision (SS) of the ICDS & Health Supervisory Cadre; Strategic Use of Data (SUD) & Convergent Action Plan; Involving Panchayati Raj Members (PRIs) for improved Co-Coverage of nutrition services; THR offering refinement; All intervention component together
  Arms: A&T- intensive

SUMMARY:
Progress on child growth outcomes such as stunting requires both direct and indirect actions across multiple sectors. Recognizing the importance of multisector approaches in reducing child undernutrition, Alive & Thrive (A&T) India aims to improve the quality of health and nutrition services, as well as their convergence at the household level with other available nutrition-sensitive services, in order to improve MIYCN behaviors, and ultimately decrease malnutrition in Gujarat. In line with government priorities, A&T designed a suite of system strengthening interventions including capacity building, supportive supervision, strategic use of data, improved food supplementation and engagement with local governance to improve the quality and co-coverage of nutrition-relevant services in three districts in Gujarat. This proposed evaluation aims to assess the feasibility of integrating multi-sectoral interventions using a cluster-randomized design with cross-sectional baseline and endline surveys.

DETAILED DESCRIPTION:
This study uses a cluster-randomized design with cross-sectional baseline and endline surveys to generate a proof-of-concept around an implementation model that aims to strengthen systems for delivery of individual interventions and to strengthen convergence of multiple interventions on the same households/families. The primary objectives of the study are to answer the following questions:

1. To what extent and through which pathways can overall system strengthening approaches improve quality of delivery of health and ICDS services?
2. To what extent and through which pathways do system strengthening approaches and focused local efforts to engage multiple sectors improve coverage of individual interventions and co-coverage of multiple interventions in the first 1,000-days?
3. Can efforts to improve the nutritional value and palatability of take-home rations within the ICDS increase acceptability and use?

This study will also measure a range of secondary outcomes, for each research question as well as outcomes that pertain to the pathways of impact of the five intervention components. These include

* MIYCN capacity building
* Strengthening Supportive Supervision (SS) of the ICDS & Health Supervisory Cadre
* Strategic Use of Data (SUD) & Convergent Action Plan
* Involving Panchayati Raj Members (PRIs) for improved Co-Coverage of nutrition services
* THR offering refinement

Prior to the baseline survey, 13 out of 26 blocks from three districts randomly allocated to receive interventions. Another 13 blocks from the same three districts were randomly allocated to the comparison groups which received standard government services. The selection of three districts was based on the discussion between A&T team and the Government of Gujarat. A team comprising of representatives from A&T, IFPRI and local government worked closely to ensure matching and comparability between the intervention and comparison blocks using a propensity score matching method prior to randomization to intervention or comparison groups.

At baseline, information related to primary and secondary outcomes will be collected, along with indicators along the pathway from program inputs to outcomes. Insights on implementation will be documented throughout the evaluation period through routine meetings with the implementation teams, field visits by the research team, review of monitoring data collected by the implementation team, and backend data from the supervisory and PRI apps. Endline will be collected after approximately one year from baseline and will use mixed methods approach wherein surveys will be conducted at the sector, village, and household levels and semi-structured interviews will be conducted with the block and district staff. In addition, observations will be conducted of interactions between supervisors and FLWs at the village level. Finally, an assessment of child growth outcomes will be conducted after exploring the availability and data quality of longitudinal data being gathered at AWCs by IIPH-G, contingent on data access and approval from the state government.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with children <2 years of age who are registered with the Anganwadi Center to receive services under the ICDS
* Pregnant women in first, second and third trimester who are registered with the Anganwadi Center to receive services under the ICDS
* Frontline health workers in the areas
* Supervisors/managers in the areas
* Key informants from the Panchayati Raj Institutions (PRI)

Exclusion Criteria:

* Women who are not currently registered with the local Anganwadi center to receive ICDS services
* Age <18
* Pregnant women with severe illness or complications
* Mothers with severely ill children
* Mental health problems that make it difficult for the respondent to answer the questions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Quality of delivery of health and nutrition interventions | During pregnancy (about 9 months)
  Proportion of beneficiaries receiving all ANC care items (weigh, blood sample taken, blood pressure measured, urine sample taken, abdomen checked),THR supplements and counseling.
Acceptability of reformulated take home ration by pregnant, lactating women and children | During pregnancy (about 9 months) and up to 24 months postpartum
  Total standardized scores of acceptability to five THR organoleptic properties (taste, smell, texture, color, difficulty of eating), with higher scores representing higher acceptability.
Use of reformulated take home ration by pregnant, lactating women and children | During pregnancy (about 9 months) and up to 24 months postpartum
  Proportion of beneficiaries who consumed THR during pregnancy, lactation or early childhood
Co-coverage of multiple interventions from across sectors | During pregnancy (about 9 months) and up to 24 months postpartum
  * For pregnant women: Proportion of pregnant women receiving at least 7 out of 14 interventions (>=4 ANC, received IFA, tetanus, weighed during ANC, breast feeding and cord counselling, received THR, health & nutrition education, mosquito net, improved sanitation, clean cooking fuel, met ASHA worker at home, met AWW at home)
  * For mothers with children <2y: Proportion of mother-child pairs receiving at least 12 out of 24 interventions (≥ 4 ANC visits, received IFA, tetanus, deworming, weighed during ANC, breastfeeding and cord-care counselling, food supplementation, health and nutrition education, mosquito net, institutional birth, postnatal care for mothers and babies, postnatal food supplementation, postnatal health and nutrition education, counselling on child growth, deworming, pediatric IFA, Vitamin A supplementation, child weighing, home visits by AWW or ASHW, HHs with improved sanitation facility and cooking fuel)

SECONDARY OUTCOMES:
MIYCN knowledge of FLWs | In the 6 months prior to interview date
  Total standardized scores of correct answers to questions related to dietary diversity, micronutrients, and child feeding, with higher scores represent higher knowledge.
Supportive supervision | In the 6 months prior to interview date
  Total standardized scores of frequency and contents discussed during supervisory visits, with higher scores representing higher supervision.
Decentralized programmatic decision-making using data | In the 6 months prior to interview date
  Proportion of supervisors and frontline workers reporting use of any data (on THR distribution, growth monitoring, home visit, IFA/Ca/vaccine stocks etc) in the last 3 months.
Panchayati Raj Members (PRI) member involvement | In the 6 months prior to interview date
  Proportion of PRI members aware of all social safety net programs, ICDS and health services
Mother IYCF knowledge and practices | During pregnancy (about 9 months) and up to 24 months postpartum
  Total standardized scores of correct answers to questions related child feeding based on 2021 WHO recommendation, with higher scores representing higher knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Phuong H Nguyen, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No